CLINICAL TRIAL: NCT04469036
Title: Improving Family-Centered Pediatric Trauma Care: The Standard of Care Versus the Virtual Pediatric Trauma Center
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 1623230
Record Dates: First submitted 2020-07-08; First posted 2020-07-13 (Actual); Results first posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2024-11

CONDITIONS: Trauma; Injuries
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Stepped-wedge
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telephone Consultation (Control) (No Intervention): Telephone consultation to a pediatric trauma specialist.
- Virtual Pediatric Trauma Center (Intervention) (Experimental): The Virtual Pediatric Trauma Center uses telehealth to consult a pediatric trauma specialist.
  Interventions: Other: Virtual Pediatric Trauma Center

INTERVENTIONS:
Other: Virtual Pediatric Trauma Center — Telehealth
  Arms: Virtual Pediatric Trauma Center (Intervention)

SUMMARY:
More than 41 million children, or 55 percent of all children in the United States, live more than 30 minutes away from a pediatric trauma center. The management of pediatric trauma requires medical expertise that is only available at Level I pediatric trauma centers, which are specialized pediatric referral hospitals located in large urban cities. Smaller hospitals lack pediatric trauma expertise and resources to properly care for these children. When a small hospital receives a child with trauma, the standard of care is to conduct a telephone consultation to a pediatric trauma specialist, err on the side of safety, and transfer the child to the regional Level I pediatric trauma center.

A newer model of care, the Virtual Pediatric Trauma Center (VPTC), uses live video, or telemedicine, to bring the expertise of a Level I pediatric trauma center virtually to patients at any hospital emergency department. While the VPTC model is being used more frequently, the advantages and disadvantages of these two systems of care remain unknown, particularly with regard to parent/family-centered outcomes.

The goal of this study is to optimize the patient and family experience and to minimize distress, healthcare utilization, and out-of-pocket costs following the injury of a child. The results of this project will help to optimize communication, confidence, and shared decision making between parents/families and clinical staff from both the transferring and receiving hospitals.

DETAILED DESCRIPTION:
The American College of Surgeons Committee on Trauma (ACS-COT) has been committed to improving the care provided to injured patients since 1922. An essential component of their efforts has been the creation of minimum standards for trauma facilities and a tiered trauma care system. As detailed in the ACS-COT published guidelines, Resources for Optimal Care of the Injured Patient, these standards outline the five levels of trauma facilities that define varying levels of commitment, readiness, resources, policies, patient care, and performance improvement. A Level I trauma center is the highest designation and is only granted to hospitals that are able to provide the highest level of care to all injured patients. The ACS-COT Trauma Center Verification process has been instrumental in improving outcomes among injured children and adults, and has become the national model of trauma care coordination as well as the prototype for trauma care on an international level.

While the regionalization of trauma care has resulted in improved outcomes, the current standard of care has created disparities in access for patients injured in geographically isolated locations. When children living in remote communities are injured and present to a non-pediatric trauma center emergency department (ED), they are transferred to the regionalized Level I pediatric trauma center. In more than half of the states in the US, a majority of children live more than 30 miles from a designated Level I pediatric trauma center. Currently, there are more than 41 million children in the US that have poor access to care, living more than 30 miles from a pediatric trauma center, and it is these children who would benefit the most from a re-engineered system of care that addresses the disparities in access for injured children.

Because the current regionalization of trauma centers has created disparities in access, many pediatric trauma experts, including health policy makers, health services researchers, and front line clinicians, have advocated for the use of telemedicine so that the Level I pediatric trauma center expertise can be transmitted to the receiving EDs where a majority of pediatric trauma patients initially present. This newer system of care has been commonly referred to as the "Virtual Pediatric Trauma Center" (VPTC) and is increasingly used by many hospitals and EDs throughout the country. The VPTC creates a model of care that connects EDs in non-Level I trauma centers using telemedicine to bring expert pediatric trauma care to the bedside of injured children, no matter which hospital the patient presents to first. While this newer model of care enables participation of parents/families in the initial trauma care, there is conflicting and limited literature comparing this model to the current standard of care as it relates to parent/family-experience and distress, healthcare utilization, and financial impact on parents/families.

As evidence, in preparation for the original proposal for this study, we conducted three meetings with community advisory boards, which laid the foundation for the study design and evaluation (see: Community and Stakeholder Involvement During Study Development below). For the resubmission of that proposal, we reconvened with members from each of these boards to focus more on parent/family-centered measures. Our team of clinical investigators, consortium hospital partners, as well as our two broadly representative community advisory boards, are confident that these two models of care can be effectively compared, and that the results will provide important solutions to problems facing families wanting to improve specialized trauma care for children. As highlighted in the PCORI Research Prioritization Topic Brief entitled, "Rural Trauma Care," improving rural trauma care is a "high-impact target."20 Recent data derived on adult patients have documented the impact that telemedicine can have on clinical outcomes in a variety of trauma settings. Having the core members of a regionalized Level I pediatric trauma center available virtually at the bedside of injured children has the potential to have a positive impact on the parent and family involvement in shared decision making, which may reduce unnecessary and financially burdensome transfers. Alternatively, parents and families may prefer to err on the side of safety and have an injured child immediately transferred to the regional Level I pediatric trauma center, so delaying or avoiding the transfer of an injured child to a better equipped and staffed facility could result in increased parent/family distress, healthcare utilization, and out-of-pocket costs. Hence, a rigorous comparison of the two prevailing models of care is needed to inform the choice between them.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients (<18 years old) with an acute injury at the time of a transfer consultation call to UC Davis Trauma Surgery, Orthopedic Surgery, or Neurosurgery from eleven outside emergency departments*
* Parents/guardians of the above patients will be contacted to complete surveys

Exclusion Criteria:

* Pediatric patients who are wards of the state
* Pediatric patients who die before the 3-day survey is administered
* Pediatric patients receiving cardiopulmonary resuscitation prior to presentation to either the outside or UC Davis emergency department

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 595 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2022-11-27 (Actual); Study Completion 2022-11-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of California-Davis, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The "Virtual Pediatric Trauma Center" (VPTC) is a model of care that utilizes telemedicine for acutely injured children presenting to non-pediatric trauma center hospitals to obtain consultations from pediatric trauma specialists. This randomized controlled trial compared the standard of care (telephone consultation from a referring non-pediatric trauma center connected to a pediatric trauma specialist at a level I pediatric trauma center) to the VPTC model of care (telemedicine consultation between the referring facility and pediatric specialist) for pediatric trauma injuries. Data comparing the two models was collected to assess parent/family experience of care and distress, transfer rates, healthcare utilization, and financial impact on parents/families. 595 children were enrolled during the two-year active study period and data was collected from parent/family surveys and the electronic health record (EHR).
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: All study data housed at the University of California Davis Health will be destroyed after seven years after completion of the study.
  Once study data has been deposited in the ICPSR repository, ICPSR will maintain the full data package following their established routine procedures for restricted-use classification.
Access Criteria: Data collected for this project includes information gathered from participant surveys and the UCDH EHR; this data will be deposited and housed in the ICPSR repository in perpetuity.
  The VPTC model of care is an innovative intervention designed to address access disparities that were exacerbated by regionalization of Level I pediatric trauma centers. The intervention leveraged telemedicine to facilitate real-time consultations and care coordination between non-pediatric emergency departments and level I pediatric trauma centers. Data from this study may be of interest to practitioners, payors, policy makers, and patients.

REFERENCES:
- [Derived] Marcin JP, Tancredi DJ, Galante JM, Rinderknecht TN, Haus BM, Leshikar HB, Zwienenberg M, Rosenthal JL, Grether-Jones KL, Hamline MY, Hoch JS, Kuppermann N. Measuring the impact of a "Virtual Pediatric Trauma Center" (VPTC) model of care using telemedicine for acutely injured children versus the standard of care: study protocol for a prospective stepped-wedge trial. Trials. 2022 Dec 27;23(1):1051. doi: 10.1186/s13063-022-06996-1. PMID 36575536

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for this project began on 11/30/2020. Electronic medical record data was collected from a Transfer Center report that included children who presented to one of the participating sites with a transfer consultation to UC Davis Trauma, Orthopedics, or Neurosurgery services.
Pre-assignment Details: We used a prospective stepped-wedge trial design. After 6-month pre-implementation, study began with all 10 hospitals beginning in standard of care and patients enrolled for 13, 8-week periods. 706 patients were assessed for eligibility, 73 patients did not meet inclusion criteria and 38 were excluded from the study. 595 enrolled patients were then randomized to the study. Parents (not enrolled in the study) of the patients were then contacted to complete surveys.
Units Other Than Participants: Hospitals
Groups:
- Virtual Pediatric Trauma Center (Intervention): The Virtual Pediatric Trauma Center uses telehealth for consultation with a pediatric trauma specialist.
- Telephone Consultation (Control): Telephone consultations uses audio-only to connect with a pediatric trauma specialist.
Period: Start of Standard of Care: 8-week Period
Arm/Group | Virtual Pediatric Trauma Center (Intervention) | Telephone Consultation (Control)
Started | 0; 0 Hospitals | 32; 10 Hospitals
Completed | 0; 0 Hospitals | 32; 10 Hospitals
Not Completed | 0; 0 Hospitals | 0; 0 Hospitals
Period: Hospital Randomization Phase 1
Arm/Group | Virtual Pediatric Trauma Center (Intervention) | Telephone Consultation (Control)
Started | 5; 1 Hospitals | 32; 9 Hospitals
Completed | 5; 1 Hospitals | 32; 9 Hospitals
Not Completed | 0; 0 Hospitals | 0; 0 Hospitals
Period: Hospital Randomization Phase 2
Arm/Group | Virtual Pediatric Trauma Center (Intervention) | Telephone Consultation (Control)
Started | 7; 2 Hospitals | 46; 8 Hospitals
Completed | 7; 2 Hospitals | 46; 8 Hospitals
Not Completed | 0; 0 Hospitals | 0; 0 Hospitals
Period: Hospital Randomization Phase 3
Arm/Group | Virtual Pediatric Trauma Center (Intervention) | Telephone Consultation (Control)
Started | 21; 3 Hospitals | 29; 7 Hospitals
Completed | 21; 3 Hospitals | 29; 7 Hospitals
Not Completed | 0; 0 Hospitals | 0; 0 Hospitals
Period: Hospital Randomization Phase 4
Arm/Group | Virtual Pediatric Trauma Center (Intervention) | Telephone Consultation (Control)
Started | 23; 4 Hospitals | 28; 6 Hospitals
Completed | 23; 4 Hospitals | 28; 6 Hospitals
Not Completed | 0; 0 Hospitals | 0; 0 Hospitals
Period: Hospital Randomization Phase 5
Arm/Group | Virtual Pediatric Trauma Center (Intervention) | Telephone Consultation (Control)
Started | 35; 5 Hospitals | 24; 5 Hospitals
Completed | 35; 5 Hospitals | 24; 5 Hospitals
Not Completed | 0; 0 Hospitals | 0; 0 Hospitals
Period: Hospital Randomization Phase 6
Arm/Group | Virtual Pediatric Trauma Center (Intervention) | Telephone Consultation (Control)
Started | 34; 6 Hospitals | 15; 4 Hospitals
Completed | 34; 6 Hospitals | 15; 4 Hospitals
Not Completed | 0; 0 Hospitals | 0; 0 Hospitals
Period: Hospital Randomization Phase 7
Arm/Group | Virtual Pediatric Trauma Center (Intervention) | Telephone Consultation (Control)
Started | 23; 7 Hospitals | 8; 3 Hospitals
Completed | 23; 7 Hospitals | 8; 3 Hospitals
Not Completed | 0; 0 Hospitals | 0; 0 Hospitals
Period: Hospital Randomization Phase 8
Arm/Group | Virtual Pediatric Trauma Center (Intervention) | Telephone Consultation (Control)
Started | 36; 8 Hospitals | 5; 2 Hospitals
Completed | 36; 8 Hospitals | 5; 2 Hospitals
Not Completed | 0; 0 Hospitals | 0; 0 Hospitals
Period: Hospital Randomization Phase 9
Arm/Group | Virtual Pediatric Trauma Center (Intervention) | Telephone Consultation (Control)
Started | 40; 9 Hospitals | 7; 1 Hospitals
Completed | 40; 9 Hospitals | 7; 1 Hospitals
Not Completed | 0; 0 Hospitals | 0; 0 Hospitals
Period: Hospital Randomization Phase 10
Arm/Group | Virtual Pediatric Trauma Center (Intervention) | Telephone Consultation (Control)
Started | 47; 10 Hospitals | 0; 0 Hospitals
Completed | 47; 10 Hospitals | 0; 0 Hospitals
Not Completed | 0; 0 Hospitals | 0; 0 Hospitals
Period: Hospital Randomization Phase 11
Arm/Group | Virtual Pediatric Trauma Center (Intervention) | Telephone Consultation (Control)
Started | 54; 10 Hospitals | 0; 0 Hospitals
Completed | 54; 10 Hospitals | 0; 0 Hospitals
Not Completed | 0; 0 Hospitals | 0; 0 Hospitals
Period: Hospital Randomization Phase 12
Arm/Group | Virtual Pediatric Trauma Center (Intervention) | Telephone Consultation (Control)
Started | 44; 10 Hospitals | 0; 0 Hospitals
Completed | 44; 10 Hospitals | 0; 0 Hospitals
Not Completed | 0; 0 Hospitals | 0; 0 Hospitals

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Virtual Pediatric Trauma Center (Intervention) | Telephone Consultation (Control) | Total
Number analyzed (Participants) | 369 | 226 | 595
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 369 | 226 | 595
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.1 (5.2) | 8 (5.1) | 8 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 142 | 81 | 223
  Male | 227 | 145 | 372
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 125 | 74 | 199
  Non-Hispanic, Black | 27 | 18 | 45
  Non-Hispanic, White | 170 | 109 | 279
  Non-Hispanic, Other | 47 | 25 | 72
Insurance Type [Count of Participants; unit: Participants]
  Commercial | 129 | 82 | 211
  Medicaid | 240 | 144 | 384
Language [Count of Participants; unit: Participants]
  English | 331 | 208 | 539
  Spanish | 23 | 15 | 38
  Other/Missing | 15 | 3 | 18
Injury Severity Score [Count of Participants; unit: Participants] — Injury Severity Scores range from 1 to 75. A score of 75 is derived from either three Abbreviated Injury Scale 5 injuries or from one Abbreviated Injury Scale 6 injury. Any Abbreviated Injury Scale 6 (maximal) injury is an automatic maximal Injury Severity Score of 75, regardless of any other injuries that may also be found.
  Data in the table represent the number of patients that scored within the respective ranges.
  Participants
    0 - 8 (minor injuries) | 290 | 159 | 449
    9 - 15 (moderate injuries) | 55 | 52 | 107
    24 (severe injuries) | 24 | 15 | 39
Glasgow Coma Scale Score [Count of Participants; unit: Participants] — A Glasgow Coma Scale (GCS) score of 15 is the best possible score, indicating that a patient is fully awake, alert, and responsive. A score of 8 or fewer usually indicates a coma, with lower scores indicating deeper comas. A score of 3 is the worst possible score, indicating that the patient is completely unresponsive. The data below indicates the number of patients that either scored 15 on the Glasgow Coma Scale, or patients that scored below 15.
  Participants
    3 - 14 | 24 | 18 | 42
    15 | 345 | 208 | 553
Distance in miles from outlying hospital [Mean (Standard Deviation); unit: Miles] | 38.2 (36.3) | 48.8 (52.4) | 42.3 (43.4)

OUTCOME MEASURES:

1. Primary Outcome: Consumer Assessment of Healthcare Providers and Systems Child Hospital Survey Communication Subscale
Description: 19 questions from the Communication with Parent Subscale of the Consumer Assessment of Healthcare Providers and Systems Child Hospital Survey. We created an "Overall" score representing the sum of the subscales. Analyses compared normalized scores (from 0 to 1) for the overall score and each of the subscale scores, which higher scores implying improved experiences of care. Adjusted mean differences were calculated using mixed-effects regression models, accounting for a small number of potential confounders, with splines to adjust for calendar time.
  We collected data on the following measures: "When your child was admitted to this emergency department" (Yes, definitely; Yes, somewhat; No), "Your experience with nurses" (Never, Sometimes, Usually, Always), "Your experience with doctors" (Never, Sometimes, Usually, Always), "Your experience with providers" (Never, Sometimes, Usually, Always), "When your child left this hospital" (Yes, definitely; Yes, somewhat; No)
Time Frame: 3 days after emergency department visit
Population: All participants who received either Virtual Pediatric Model of Care or a Telephone Consultation that reported Consumer Assessment of Healthcare Providers and Systems Child Hospital Survey scores, data analyzed as Intention-to-Treat.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual Pediatric Trauma Center (Intervention) | Telephone Consultation (Control)
Number analyzed (Participants) | 199 | 146
score on a scale
  Overall patient experience of care | 0.769 (0.209) | 0.775 (0.223)
  When Your Child Was Admitted to this Hospital | 0.735 (0.335) | 0.747 (0.357)
  Your Experience with Nurses at [hospital name] | 0.878 (0.205) | 0.890 (0.214)
  Your Experience with Doctors at [hospital name] | 0.872 (0.230) | 0.865 (0.254)
  Your Experience with Providers at [hospital name] | 0.859 (0.208) | 0.875 (0.203)
  When Your Child Left the ED at [hospital name] | 0.645 (0.331) | 0.632 (0.359)

2. Primary Outcome: 3-Day State-Trait Anxiety Inventory Form Y
Description: State-Trait Anxiety Inventory measures state anxiety levels in adults. Responses for the State Anxiety scale assess intensity of current feelings "at this moment". Participant response choices include: 1) not at all, 2) somewhat, 3) moderately so, and 4) very much so. Data below represent total mean and standard deviation scores between the two groups.
Time Frame: 3 days after emergency department visit
Population: All participants who received either Virtual Pediatric Model of Care or a Telephone Consultation that reported State-trait anxiety scores at 3-days, data analyzed as Intention-to-Treat.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual Pediatric Trauma Center (Intervention) | Telephone Consultation (Control)
Number analyzed (Participants) | 194 | 142
score on a scale | 1.775 (0.594) | 1.812 (0.620)

3. Secondary Outcome: Transfer Rates
Description: Transfer rates from the referring emergency department to the trauma center will be compared between the control and intervention groups.
Time Frame: Transfer from initial ED visit to UCDH
Population: 338 patients transferred to UC Davis Health, numbers reported in the table indicate patient disposition from UC Davis Health Emergency Department, data was analyzed using Intention-to-Treat analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Virtual Pediatric Trauma Center (Intervention) | Telephone Consultation (Control)
Number analyzed (Participants) | 369 | 226
Participants
  Transferred to UCDH | 338 | 212
  Discharged Home from UCDH ED | 127 | 73
  Admitted to the Ward | 107 | 71
  Admitted to the ICU | 32 | 32
  Taken to Operating Room | 72 | 36

4. Secondary Outcome: 30-Day Healthcare Utilization
Description: Healthcare utilization included hospitalization and re-hospitalization as measures. Two analyses were done to study 30-day healthcare utilization comparing the intervention and control group.
  First, the VPTC model of care was compared to the standard of care with respect to ED and hospital use, including transfer and subsequent care needed following initial injury. Second, the VPTC model of care was compared to the standard of care with respect to healthcare (hospital) charges.
Time Frame: 30 days after emergency department visit
Population: Healthcare Utilization of patients evaluated at 30-days after discharge following an ER visit, Intention-to-Treat analysis used.
Measure: Mean (Standard Deviation); unit: Dollars
Arm/Group | Virtual Pediatric Trauma Center (Intervention) | Telephone Consultation (Control)
Number analyzed (Participants) | 369 | 226
Dollars
  Total Post-Transfer Initial Care Charges in Dollars | 77,805 (93,219) | 79,468 (103,570)
  Total Subsequent Care Charges in Dollars | 3,228 (37,330) | 976 (8,495)
  Total 30-Day Charges in Dollars | 81,032 (105,762) | 90,443 (104,401)

5. Secondary Outcome: 3-Day Out-of-Pocket Costs
Description: At 3-days, surveys requested parents of patients to self-report medical and non-medical Out-of-Pocket costs following their ED visit.
Time Frame: 3 days after emergency department visit
Population: Modified Intention-to-Treat analysis of patients that reported 3-day Out-of-Pocket cost data.
Measure: Mean (Standard Deviation); unit: Dollars
Arm/Group | Virtual Pediatric Trauma Center (Intervention) | Telephone Consultation (Control)
Number analyzed (Participants) | 173 | 127
Dollars
  3-Day Medical Out-of-Pocket Costs in Dollars | 151 (1,521) | 507 (4,478)
  3-Day Non-Medical Out-of-Pocket Costs in Dollars | 228 (405) | 335 (735)
  3-Day Total Out-of-Pocket Costs in Dollars | 379 (1,572) | 842 (4,596)

6. Secondary Outcome: 30-Day Out-of-Pocket Costs
Description: At 30-days, surveys requested parents of patients to self-report medical and non-medical Out-of-Pocket costs following their ED visit.
Time Frame: 30 days after emergency department visit
Population: Modified Intention-to-Treat analysis of patients that reported 30-day out of pocket cost data.
Measure: Mean (Standard Deviation); unit: Dollars
Arm/Group | Virtual Pediatric Trauma Center (Intervention) | Telephone Consultation (Control)
Number analyzed (Participants) | 166 | 120
Dollars
  30-Day Medical Out-of-Pocket Costs in Dollars | 247 (926) | 3,293 (31,945)
  30-Day Non-Medical Out-of-Pocket Costs in Dollars | 625 (4,670) | 216 (411)
  30-Day Total Out-of-Pocket Costs in Dollars | 872 (4,747) | 3,509 (32,022)

7. Secondary Outcome: 30-Day State-Trait Anxiety Inventory Form Y
Description: State-Trait Anxiety Inventory was used to measure state anxiety levels. Responses for the State Anxiety scale assess intensity of current feelings "at this moment". Participant choices included: 1) not at all, 2) somewhat, 3) moderately so, and 4) very much so. Data below represent total mean and standard deviation scores between the two groups.
Time Frame: 30 days after emergency department visit using Intention-to-Treat analysis.
Population: All participants who received either Virtual Pediatric Model of Care or a Telephone Consultation that reported State-trait anxiety scores at 30-days, data analyzed as Intention-to-Treat.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Virtual Pediatric Trauma Center (Intervention) | Telephone Consultation (Control)
Number analyzed (Participants) | 190 | 134
score on a scale | 1.776 (0.647) | 1.798 (0.621)

ADVERSE EVENTS:
Time Frame: 2 years
Groups:
- Virtual Pediatric Trauma Center: The Virtual Pediatric Trauma Center (VPTC), uses live video, or telehealth, to bring the expertise of a Level I pediatric trauma center virtually to patients at a hospital emergency department.
  Virtual Pediatric Trauma Center: Telehealth
- Telephone Consultation: Telephone consultation to a pediatric trauma specialist
Arm/Group | Virtual Pediatric Trauma Center | Telephone Consultation
All-Cause Mortality (participants affected / at risk) | 0/369 | 0/226
Serious Adverse Events (participants affected / at risk) | 0/369 | 0/226
Other Adverse Events (participants affected / at risk) | 0/369 | 0/226

LIMITATIONS AND CAVEATS:
* Expanding the existing clinical workflow to conduct telehealth visits was not universally supported given the limited physician staff.
* Intervention intended to inform clinical-decision making, but was adapted towards supporting parents. Nurse practitioners became the primary initiator of consultations instead of the trauma surgeons.
* Partner sites had more unique needs and workflows as the program was expanding, requiring unique solutions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-22): https://cdn.clinicaltrials.gov/large-docs/36/NCT04469036/Prot_SAP_000.pdf